CLINICAL TRIAL: NCT01581398
Title: A Phase 3, Randomized, Multi-center, Active-Controlled, Open-label Study to Evaluate the Efficacy and Safety of Peginterferon Alfa-2b (40kD, Y Shape) in Combination With Ribavirin in Chinese Chronic Hepatitis C Patients
Brief Title: Efficacy and Safety Study of Peginterferon Alfa-2b in Chinese Chronic Hepatitis C Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TB1203IFN
Record Dates: First submitted 2012-02-16; First posted 2012-04-20 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Hepatitis C
Keywords: Peginterferon; Pegasys; Sustained virus response; HCV
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A1(Genotype2/3) (Experimental): Ypeginterferon alfa-2b 180μg/week, in combination with Ribavirin 800mg/day
  Interventions: Drug: Ypeginterferon alfa-2b
- A2(Genotype 2/3) (Active Comparator): Pegasys 180μg/week, in combination with Ribavirin 800mg/day
  Interventions: Drug: Pegasys
- B1(Non-genotype 2/3) (Experimental): Ypeginterferon alfa-2b 180μg/week, in combination with Ribavirin 1000-1200mg/day based on body weight
  Interventions: Drug: Ypeginterferon alfa-2b
- B2(Non-genotype 2/3) (Active Comparator): Pegasys 180μg/week, in combination with Ribavirin 1000-1200mg/day based on body weight.
  Interventions: Drug: Pegasys

INTERVENTIONS:
Drug: Ypeginterferon alfa-2b — sc, qw, 24 weeks.
  Arms: A1(Genotype2/3)
Drug: Pegasys — sc, qw, 24 weeks.
  Arms: A2(Genotype 2/3)
Drug: Ypeginterferon alfa-2b — sc, qw, 48 weeks.
  Arms: B1(Non-genotype 2/3)
Drug: Pegasys — sc, qw, 48 weeks.
  Arms: B2(Non-genotype 2/3)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Peginterferon alfa-2b (40KD, Y shape, the followings will refer as Ypeginterferon alfa-2b for short), at a dose of 180μg/week, in combination with Ribavirin in Chinese chronic hepatitis C patients. The study will first group patients into two sub-study, genotype 2/3 and non-genotype 2/3, depending on the HCV genotype that infected. In the genotype 2/3 sub-study about 219 patients will be enrolled, and eligible patients are randomized at 2:1 ratio into Ypeginterferon alfa-2b group or active control group (Pegasys), receiving 24 weeks of interferon therapy and oral daily Ribavirin at a dose of 800mg/d. In the non-genotype 2/3 sub-study about 507 patients will be enrolled, and eligible patients are randomized at 2:1 ratio into Ypeginterferon alfa-2b group or active control group (Pegasys), receiving 48 weeks of interferon therapy and oral daily Ribavirin 1000-1200mg/day , basing on body weight. All patients will be followed for 24 weeks after the end of therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18~65 years
* Hepatitis virus C chronic infection evidences: HCV RNA or anti-HCV positive>6 months,or other evidences supporting diagnosis of chronic hepatitis C infection
* HCV RNA≥2000IU/mL, anti-HCV positive at screening
* Pregnancy tests for female patients must be negative. All patients must take effective contraception measures during the study period
* Signed informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Mental or psychology disorder
* ANC<1500/mm3, or PLT<90,000/mm3, or Hb<ULN(Upper limit of Normal)
* Received interferon treatment within the previous 6 months or shown no-response to previous interferon treatment
* Co-infection with HIV, HAV, HBV, HEV
* Evidence of hepatic decompensation (e.g: Child Plug≥B, prothrombin time prolonged more than 3 seconds, TBil>2ULN, Alb<35g/L)
* Hepatocarcinoma or suffering from any other malignant tumor
* Not well controlled endocrine diseases(e.g:thyroid disfunction, mellitus mellitus)
* Significant function damage in any major organs (e.g: heart, lung, kidney)
* Involved in other investigation within the previous 3 months
* Other conditions which in the opinion of the investigator precluding enrollment into the study (e.g: poor compliance)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with sustained virologic response (defined as HCV RNA<15IU/ml at 24 weeks after the end of therapy) | 24 weeks after the end of therapy

SECONDARY OUTCOMES:
Proportion of patients with HCV RNA undetectable (defined as HCV RNA <15IU/ml) | at weeks 4, 12, 24 for genotype 2/3, and weeks 4, 12, 24 and 48 for non-genotype 2/3

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lai, MD, PhD, Principal Investigator — Peking University People's Hospital
Locations (42):
- China (42):
  - 302 Military Hospital, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - Beijing Youyi Hospital, capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - First Affiliated Hospital of Jilin University, Changchun
  - Xiangya Hospital, Central-south University, Changsha
  - Xiangya Second Hospital, Central-south University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Second Affiliated Hospital Chongqing Medical University, Chongqing
  - Southwest Hospital, Chongqing
  - Fuzhou Infectious Disease Hospital, Fuzhou
  - Guangzhou Eighth People's Hospital, Guangzhou
  - Nanfang Hospital, Guangzhou
  - Third Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - First Affiliated Hospital of Guangxi Medical University, Guilin
  - Affiliated Hospital of Guiyang Medical College, Guiyang
  - First Affiliated Hospital, Zhejiang University, Hangzhou
  - Second Affiliated Hospital of Harbin Medical University, Harbin
  - First Affiliated Hospital of Anhui Medical University, Hefei
  - Jinan Infectious Disease Hospital, Jinan
  - First Affiliated Hospital of Lanzhou University, Lanzhou
  - First Affiliated Hospital of Nanchang University, Nanchang
  - 81 Military Hospital, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Second Hospital of Nanjing, Nanjing
  - 85 Militay Hospital, Shanghai
  - Huashan Hospital, Shanghai
  - Renji Hospital, Shanghai
  - Ruijing Hospital, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - Third Affiliated Hospital, Hebei Medical University, Shijiazhuang
  - First Affiliated Hospital, Shanxi University, Taiyuan
  - Tianjin Third Central Hospital, Tianjin
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Tangdu Hospital, Fourth Military Medical University, Xi'an
  - Xijing Hospital, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Hennan Provincial People's Hospital, Zhengzhou